CLINICAL TRIAL: NCT06885073
Title: Non-invasive Central Venous Pressure Estimation in Pediatric Patients
Acronym: CPMX-CVP-Ped
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Compremium AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CPMX-CVP-Ped
Record Dates: First submitted 2025-03-04; First posted 2025-03-20 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Central Venous Pressure
Keywords: central venous pressure; venous hypertension

STUDY DESIGN:
Masking Description: The investigator performing the measurement with CPMX2 is blinded to the invasive CVP measurement until the assessment is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- CPMX2 measurement arm (Experimental): CPMX2 measurements will be compared against invasive CVP measurements
  Interventions: Device: CPMX2

INTERVENTIONS:
Device: CPMX2 — CPMX2 - Non-invasive pressure estimation

SUMMARY:
Central Venous Pressure (CVP) is a standard parameter for hemodynamic monitoring and is currently measured through the insertion of a catheter. The pediatric population is especially vulnerable to risks associated to this invasive procedure, including infection, thrombosis, and pneumothorax. The proposed pilot study will evaluate safety and preliminary efficacy of a new non-invasive ultrasound-based venous occlusion pressure (VOP) monitoring device (CPMX2) in children equipped with an invasive catheter for CVP monitoring as part of standard of care.

ELIGIBILITY:
Inclusion Criteria

* Provision of signed and dated informed consent form
* Male or female
* Age: birth to 21 years of age
* Equipped with a central venous catheter (CVC) for central venous pressure (CVP) monitoring indication as part of standard of care, or undergoing cardiac catheterization.

Exclusion Criteria:

* Weight less than 2.5kg at the time of enrollment.
* Bilateral external jugular veins not accessible due to vascular access or dressing.
* Bilateral skin lesion contraindicating neck Ultrasound
* Active bleeding
* Clinically unstable, per clinical assessment by attending physician and/or surgeon

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety of external jugular venous occlusion pressure measured non-invasively with CPMX2 to estimate CVP in pediatric patients. | Up to 4 days
  Safety: Safety of the device shall be evaluated by systematically reporting DDs, ADEs and SADEs and by monitoring the frequency and incidence of these events. The practitioner will be asked to identify any new risks arising during the measurements using the investigational device.

OTHER OUTCOMES:
Preliminary accuracy of external jugular venous occlusion pressure measured with CPMX2 to estimate CVP | Up to 4 days
  Preliminary accuracy: Accuracy of external jugular venous occlusion pressure measured with CPMX2 to estimate CVP will be evaluated against concomitant invasive CVP measurement with the standard of care catheter by computing the correlation coefficient and Bland-Altman analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thalhammer C, Aschwanden M, Jaeger KA. Letter by Thalhammer et al regarding article, "External carotid artery-internal jugular vein fistula: a complication of internal jugular cannulation". Circulation. 2006 Sep 26;114(13):e517; author reply e518. doi: 10.1161/CIRCULATIONAHA.106.636571. No abstract available. PMID 17000916